CLINICAL TRIAL: NCT00356889
Title: A Phase II Trial of Bevacizumab and Erlotinib in Patients With Advanced Biliary Tumors
Brief Title: Bevacizumab and Erlotinib Hydrochloride in Treating Patients With Metastatic or Unresectable Biliary Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00115; MC044G; CDR0000484566 (Registry Identifier: PDQ (Physician Data Query)); N01CM17104 (NIH); NCT01646957 (obsolete NCT alias); NCT01664416 (obsolete NCT alias)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-04

CONDITIONS: Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Gastrointestinal Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and Erlotinib Hydrochloride (Experimental): Patients receive 5 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15 and 150 mg oral erlotinib hydrochloride daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Tumor tissue and blood specimens are collected periodically for correlative studies. Specimens are examined by immunohistochemistry for epidermal growth factor receptor (EGFR) and P-EGFR protein levels; AKT p-AKT, mitogen-activated protein kinase (MAPK) and P-MAPK protein levels; and vascular endothelial growth factor receptor (VEGFR)-1 and VEGFR-2 protein levels. EGFR mutations are detected by laser capture microdissection. Enzyme-linked immunosorbent assay is used to measure total and free serum VEGF levels.
  Interventions: Drug: erlotinib hydrochloride; Biological: bevacizumab

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally, 150 mg, once daily.
  Other Names: CP-358,774; erlotinib; OSI-774
Biological: bevacizumab — Given IV, 5mg/kg on days 1 and 15 every cycle
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with erlotinib hydrochloride works in treating patients with metastatic or unresectable biliary tumors. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab and erlotinib hydrochloride may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving bevacizumab together with erlotinib hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the objective response rate in patients with metastatic or unresectable cholangiocarcinoma treated with bevacizumab and erlotinib hydrochloride.

SECONDARY OBJECTIVES:

I. Evaluate time to progression in these patients.

II. Evaluate overall and progression-free survival of these patients.

III. Evaluate the adverse events associated with this regimen. OUTLINE: This is an open-label, multicenter study.

Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Criteria:

* Absolute neutrophil count >= 1,500/mm3
* Histologically or cytologically confirmed cholangiocarcinoma or gallbladder carcinoma:

  * Metastatic or surgically unresectable disease
* Measurable disease, defined as >= 1 lesion whose longest diameter can be accurately measured as >= 2.0 cm with conventional techniques or as > 1.0 cm with spiral CT scan:

  * Spiral CT scan imaging must be used for pre- and post-treatment tumor measurements of lesions measuring >= 1.0 cm to < 2.0 cm
* Clinical lesions will only be considered measurable when they are superficial

  * Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung
* No ampulla of Vater tumors
* No evidence of CNS disease
* Life expectancy >= 3 months
* ECOG performance status 0-2
* Platelet count >= 75,000/mm3
* Total bilirubin =< 2 times ULN
* ALT and AST =< 2.5 times ULN
* Creatinine =< 2 mg/dL
* Albumin >= 2.5 g/dL
* Alkaline phosphatase =< 5 times ULN
* Urine protein:creatinine ratio < 1.0 OR 24-hour urine protein < 1000 mg
* No concurrent illness or medical condition, including any of the following:

  * Impairment of gastrointestinal (GI) function or disease that may significantly alter the absorption of erlotinib hydrochloride
  * Requirement for IV alimentation
* No concurrent illness or medical condition, including any of the following:

  * Active peptic ulcer disease;
  * Serious or nonhealing wound, ulcer, or bone fracture;
  * GI bleed that required procedural intervention within the past 3 months
* No concurrent illness or medical condition, including any of the following:

  * Abdominal fistula, GI perforation, or intra-abdominal abscess within the past 28 days
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Psychiatric illness or social situation that would limit study compliance
* No other malignancy within the past 3 years
* No abnormalities of the cornea
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No clinically significant cardiovascular disease
* More than 4 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* No significant traumatic injury within the past 28 days
* No prior systemic anticancer therapy for metastatic gallbladder or bile duct cancer
* More than 28 days since prior major surgery [Note: Insertion of a vascular access device is not considered major/minor surgery]
* More than 2 weeks since prior minor surgery [Note: Insertion of a vascular access device is not considered major/minor surgery]
* More than 7 days since prior core biopsy
* No concurrent major surgery
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any other therapy or supportive care considered investigational
* No concurrent enzyme-inducing antiepileptic drugs or any other CYP3A4 inducer, such as rifampin or Hypericum perforatum
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents or other concurrent anticancer therapies
* No concurrent prophylactic hematopoietic colony-stimulating factors
* Concurrent full-dose anticoagulants allowed provided PT/INR is > 1.5 and both of the following criteria are met:

  * In-range INR on a stable dose of oral anticoagulant OR on a stable dose of low molecular weight heparin
* AND (continued from above) No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels, gastrointestinal ulcerations, or known varices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-six patients were enrolled between August 2006 and April 2008 at eight sites in the Phase II Consortium. The data are reported as of November 2009.
Pre-assignment Details: Three patients were ineligible after starting treatment (brain metastases, alteration in diagnosis, colitis). Two of these participants reported adverse events. Therefore, 56 participants were used for baseline, 53 patients were used for endpoint analyses, and 55 participants were used to report toxicity.
Groups:
- Bevacizumab and Erlotinib Hydrochloride: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
  Tumor tissue and blood specimens are collected periodically for correlative studies. Specimens are examined by immunohistochemistry for epidermal growth factor receptor (EGFR) and P-EGFR protein levels; AKT p-AKT, mitogen-activated protein kinase (MAPK) and P-MAPK protein levels; and vascular endothelial growth factor receptor (VEGFR)-1 and VEGFR-2 protein levels. EGFR mutations are detected by laser capture microdissection. Enzyme-linked immunosorbent assay is used to measure total and free serum VEGF levels.
Period: Overall Study
Arm/Group | Bevacizumab and Erlotinib Hydrochloride
Started | 56
Completed | 53
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Erlotinib Hydrochloride
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 63.5 [31 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 50
  Australia | 2
  Singapore | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Confirmed Tumor Responses.
Description: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the target lesions.
  A confirmed tumor response is defined to be either a Complete Response or a Partial Response noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. Confirmed tumor responses will be evaluated using the first 6 cycles of treatment. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment and had one post-baseline disease assessment will be evaluable for response. Forty-nine of the 53 eligible patients had at least one post-baseline disease assessment and were evaluable for this endpoint.
Time Frame: After 6 courses of treatment. Each course lasts 28 days.
Measure: Number; unit: participants
Groups:
- Bevacizumab and Erlotinib Hydrochloride: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride daily on days 1-28. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.
Arm/Group | Bevacizumab and Erlotinib Hydrochloride
Number analyzed (Participants) | 49
participants
  Partial Response (PR) | 6
  Complete Response (CR) | 0

2. Secondary Outcome: Survival Time
Description: Estimated using the method of Kaplan-Meier (1958).
Time Frame: From registration to death due to any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab and Erlotinib Hydrochloride
Number analyzed (Participants) | 53
months | 9.9 [7.2 to 13.6]

3. Secondary Outcome: Time to Disease Progression
Description: Estimated using the method of Kaplan-Meier (1958).
Time Frame: From registration to documentation of disease progression, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab and Erlotinib Hydrochloride
Number analyzed (Participants) | 53
months | 4.4 [3.0 to 7.8]

4. Secondary Outcome: Duration of Response
Description: Point estimates and 95% confidence intervals were calculated using the method of Duffy and Santner (1987).
Time Frame: From the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented, assessed up to 3 years
Population: There were 6 patients with a confirmed Partial Response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab and Erlotinib Hydrochloride
Number analyzed (Participants) | 6
months | 8.4 [6.0 to 11.7]

ADVERSE EVENTS:
Arm/Group | Bevacizumab and Erlotinib Hydrochloride
Serious Adverse Events (participants affected / at risk) | 22/55
Other Adverse Events (participants affected / at risk) | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Erlotinib Hydrochloride (N=55)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 3 (3)
Infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Erlotinib Hydrochloride (N=55)
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 (28)
Hemolysis (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (2)
Dry eye syndrome (Eye disorders) | 2 (3)
Eye disorder (Eye disorders) | 3 (7)
Keratitis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (2)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 13 (25)
Anal pain (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (27)
Diarrhea (Gastrointestinal disorders) | 24 (106)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastic fistula (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 14 (18)
Nausea (Gastrointestinal disorders) | 17 (43)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 8 (12)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 3 (5)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 32 (137)
Fever (General disorders) | 2 (2)
General symptom (General disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Gallbladder infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 11 (17)
Alkaline phosphatase increased (Investigations) | 11 (29)
Aspartate aminotransferase increased (Investigations) | 16 (26)
Blood bilirubin increased (Investigations) | 16 (20)
Creatinine increased (Investigations) | 2 (2)
Leukocyte count decreased (Investigations) | 5 (8)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 8 (52)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 11 (17)
Anorexia (Metabolism and nutrition disorders) | 21 (45)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (18)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Serum albumin decreased (Metabolism and nutrition disorders) | 11 (24)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (8)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (8)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 5 (14)
Headache (Nervous system disorders) | 5 (5)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 3 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (8)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (5)
Insomnia (Psychiatric disorders) | 3 (9)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 5 (7)
Urogenital disorder (Renal and urinary disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (49)
Dry skin (Skin and subcutaneous tissue disorders) | 16 (51)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 7 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (16)
Rash desquamating (Skin and subcutaneous tissue disorders) | 42 (203)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 16 (45)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less